CLINICAL TRIAL: NCT05883319
Title: The Effect Of Cervical Mobilization And Clinical Pilates Exercises On Pain, Muscle Hardness, Head-Neck Blood Flow in Cervicogenic Headache
Brief Title: The Effect Of Cervical Mobilization And Clinical Pilates in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Uzun (Other)
Responsible Party: Sponsor-Investigator, Meltem Uzun, Director, Sanko University
Organization: Sanko University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SankoMU
Record Dates: First submitted 2022-03-22; First posted 2023-05-31 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Headache, Cervicogenic; Exercise; Therapeutics
Keywords: Cervicogenic Headache,; Pilates based exercises; Cervical mobilization; Blood flow; posture; muscle stifness
MeSH Terms: conditions — Post-Traumatic Headache; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cervical mobilization (Active Comparator): Cervical mobilization methods will be applied to 1st group for 3 days / week for 6 weeks.
  Interventions: Other: manuel therapy
- clinical pilates exercises (Active Comparator): clinical pilates exercises will be applied to 2nd group,for 3 days / week for 6 weeks.
  Interventions: Other: exercises
- cervical mobilization and clinical pilates exercises (Active Comparator): cervical mobilization and clinical pilates exercises will be applied to 3rd group,for 3 days / week for 6 weeks.
  Interventions: Other: manuel therapy; Other: exercises

INTERVENTIONS:
Other: manuel therapy — approaches will be applied for 3 days / week for 6 weeks.
  Other Names: cervical mobilization
  Arms: cervical mobilization; cervical mobilization and clinical pilates exercises
Other: exercises — approaches will be applied for 3 days / week for 6 weeks.
  Other Names: clinical pilates exercises
  Arms: cervical mobilization and clinical pilates exercises; clinical pilates exercises

SUMMARY:
Cervicogenic headache (CH) arises from cervical region problems. Various physiotherapy methods such as manual therapy approaches and exercise training are used in the treatment of CH. The aim of our study is to investigate cervical mobilization and clinical Pilates exercises on pain, muscle stiffness, head and neck blood flow in CH. Including individuals diagnosed with CH in the study. Those to be included in the study will be divided into 3 groups by a simple method. Demographic information of the individuals, age, height, weight, Body Mass Index (BMI), gender, educational status, occupation, marital status, smoking, alcohol use will be recorded. In evaluations about pain before treatment; pain intensity, pain frequency, duration and characteristics will be evaluated with Visual Analog Scale (VAS). In addition, analgesic use (frequency, amount) in headache situations will be recorded. Migraine Disability Assessment Scale (MIDAS) will be used to determine the effect of headache on quality of life. Disability Index will be used in the assessment of functional desire, and Postur Screen mobile application will be used in the assessment of posture. Range of motion(ROM) of all neck joint movements will be evaluated by CROM goniometer, deep neck flexor muscle strength by Pressure Biofeedback Unit (PBU), sternocleidomastoid(SKM), suboccipital and upper trapezius muscle stiffness myotonometer, and head-neck artery flow volume will be evaluated by Doppler ultrasound. Cervical mobilization methods will be applied to the 1st group, clinical pilates applications to the 2nd group, clinical pilates with cervical mobilization will be applied to the 3rd group for 3 days / week for 6 weeks. All evaluations were completed again after the 3rd week and after the treatment. After the obtained results are obtained, the literature will be discussed.

DETAILED DESCRIPTION:
The scope of the study, including patients over 18 years of age who applied to the Neurology outpatient clinic of Sani Konukoğlu Application and Research Hospital and presented with cervicogenic headache by a specialist. The sometimes headache frequency variable in the reference result was 5% Power analysis calculated 9 patients per group. It was decided to recruit 15 patients for the group. Inclusion criteria: CH was diagnosed, aged 18-65, had not received medical (except analgesic) treatment or physiotherapy for CH in the previous few months. Exclusion criteria: Individuals who have undergone CH surgery, history of serious heart or surgery, history of ongoing malignancy, diagnosed with epilepsy. Individuals for whom the Voluntary Consent form will be obtained will be randomly divided into groups using the minimalization method given age, gender and duration of illness.Patients will be asked not to use analgesics as much as possible during the treatment period. In the case of analgesic use, the amount and frequency will be recorded. The change in the frequency of analgesic use will also be used to evaluate the effectiveness of the applications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cervicogenic Headache
* aged 18-65
* did not receive medical (except analgesic) treatment or physiotherapy for bit Cervicogenic Headache in the previous few months

Exclusion Criteria:

* Individuals who have undergone Cervicogenic Headache surgery
* have had a serious cardiac history or surgery
* a history of ongoing or previous malignancy
* a diagnosis of epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Change of headache | 6 week
  headache intensity by Visual Analogue Scale , headache frequency and analgesic intake
Change of muscle stiffness degree | 6 week
  SKM,suboccipital and upper trapezoidal muscle stiffness with Myoton Pro
Change of blood flow degree | 6 week
  head-neck artery flow Doppler Ultrasound (US)
change of posture | 6 week
  The PostureScreen Mobile® application

SECONDARY OUTCOMES:
neck range of motion | 6 week
  range of motion by Cervical Range of Motion device
deep neck flexor muscle endurance | 6 week
  muscle endurance by Pressure Biofeedback Unit
headache life quality | 6 week
  Migraine Disability Assessment Scale for headache on quality of life.
neck functional status | 6 week
  Neck Disability Index for functional status

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Uzun, PhD(c), Study Director — Sanko University
Locations (1):
- SANKO University, Gaziantep, Please Select, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No